CLINICAL TRIAL: NCT04499365
Title: 68Ga-DOTA/NOTA-FAPI-04 PET/CT in Patients With Various Types of Cancer
Brief Title: 68Ga-FAPI PET/CT in Patients With Various Types of Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian3
Record Dates: First submitted 2020-08-01; First posted 2020-08-05 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Tumor; Positron-Emission Tomography; Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: 68Ga-DOTA/NOTA-FAPI-04 (Experimental): Each subject receive a single intravenous injection of 68Ga-DOTA/NOTA-FAPI-04, and undergo PET/CT imaging within the specificed time.
  Interventions: Drug: 68Ga-DOTA/NOTA-FAPI-04; Diagnostic Test: PET/CT scan

INTERVENTIONS:
Drug: 68Ga-DOTA/NOTA-FAPI-04 — Each patient receive a single intravenous injection of 68Ga-DOTA/NOTA-FAPI-04, and undergo PET/CT scan within specified time.
Diagnostic Test: PET/CT scan — PET/CT scan

SUMMARY:
To evaluate the potential usefulness of 68Ga-DOTA/NOTA-FAPI-04 positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various types of cancer.

DETAILED DESCRIPTION:
Subjects with various types of cancer underwent 68Ga-DOTA/NOTA-FAPI-04 PET/CT either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 68Ga-DOTA/NOTA-FAPI-04 PET/CT were calculated.

ELIGIBILITY:
Inclusion Criteria:

* (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled 68Ga-DOTA/NOTA-FAPI-04 PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant lesions; (ii) patients with pregnancy; (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 68Ga-DOTA/NOTA-FAPI-04 for each target lesion of subject or suspected primary tumor or/and metastasis.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of 68Ga-DOTA/NOTA-FAPI-04 PET/CT were calculated.
Diagnostic efficacy | 30 days
  The positive predictive value (PPV), negative predictive value (NPV)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng S, Lin J, Zhu Y, Chen Y, Zhang J, Chen X, Miao W. 68Ga-FAPI Versus 18F-FDG PET/CT in Evaluating Newly Diagnosed Breast Cancer Patients: A Head-to-Head Comparative Study. Clin Nucl Med. 2023 Mar 1;48(3):e104-e109. doi: 10.1097/RLU.0000000000004523. Epub 2023 Jan 10. PMID 36723892
- [Derived] Chen Y, Zheng S, Zhang J, Yao S, Miao W. 68Ga-DOTA-FAPI-04 PET/CT imaging in radioiodine-refractory differentiated thyroid cancer (RR-DTC) patients. Ann Nucl Med. 2022 Jul;36(7):610-622. doi: 10.1007/s12149-022-01742-8. Epub 2022 May 12. PMID 35551610
- [Derived] Zheng S, Lin R, Chen S, Zheng J, Lin Z, Zhang Y, Xue Q, Chen Y, Zhang J, Lin K, You X, Yao S, Miao W. Characterization of the benign lesions with increased 68Ga-FAPI-04 uptake in PET/CT. Ann Nucl Med. 2021 Dec;35(12):1312-1320. doi: 10.1007/s12149-021-01673-w. Epub 2021 Aug 23. PMID 34424505